CLINICAL TRIAL: NCT07183436
Title: Efficacy of Combined Intra-Articular Hyaluronic Acid and Ketorolac Versus Ketorolac Alone in the Treatment of Adhesive Capsulitis: A Randomized Controlled Trial
Brief Title: Intra-articular Corticosteroids Are Widely Used for Adhesive Capsulitis, But Alternatives Are Required for Patients With Contraindications. Hyaluronic Acid (HA) and Ketorolac Have Shown Individual Benefits. However, Evidence on Their Combination Remains Limited.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2023/497
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: Adhesive capsulitis; Frozen shoulder; Shoulder pain; Hyaluronic acid; Ketorolac; Intra-articular injection; Randomized controlled trial; Range of motion
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Hyaluronic Acid; Ketorolac

STUDY DESIGN:
Intervention Model Description: Participants randomized in a 1:1 ratio to receive either intra-articular HA+ketorolac or ketorolac alone, each followed by standardized rehabilitation
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic Acid and Ketorolac injection (Experimental): Participants received a single intra-articular injection of Hyaluronic Acid and Ketorolac
  Interventions: Drug: Intra-articular Hyaluronic Acid and Ketorolac
- Ketorolac injection (Active Comparator): Participants received a single intra-articular injection of ketorolac
  Interventions: Drug: Intra-articular Ketorolac

INTERVENTIONS:
Drug: Intra-articular Hyaluronic Acid and Ketorolac — Single intra-articular injection containing 2 mL moderate-molecular-weight hyaluronic acid (20 mg/2 mL), 1 mL ketorolac (30 mg/mL), and 2 mL lidocaine (10 mg/mL), total volume 5 mL. Administered under aseptic technique (ultrasound-guided or landmark-based) followed by standardized rehabilitation program.
  Other Names: Hyaluronic Acid and Ketorolac injection
  Arms: Hyaluronic Acid and Ketorolac injection
Drug: Intra-articular Ketorolac — single intra-articular injection containing 1 mL ketorolac (30 mg/mL), 2 mL lidocaine (10 mg/mL), and 2 mL normal saline, total volume 5 mL. Administered under aseptic technique (ultrasound-guided or landmark-based) followed by standardized rehabilitation program.
  Other Names: Ketorolac injection
  Arms: Ketorolac injection

SUMMARY:
This randomized, double-blind trial compared a single intra-articular injection of moderate-molecular-weight hyaluronic acid (HA) plus ketorolac with ketorolac alone in patients with adhesive capsulitis. Fifty-six participants were randomized into two equal groups and followed for 24 weeks. The primary outcome was shoulder function measured by the Thai Shoulder Pain and Disability Index (SPADI). Secondary outcomes included pain (VAS), passive range of motion (PROM), analgesic use, and adverse events. Both groups showed significant improvement in pain and function with no between-group difference in SPADI or VAS. The HA+ketorolac group demonstrated small but significant gains in external rotation and adduction. Both treatments were safe and well tolerated.

DETAILED DESCRIPTION:
Adhesive capsulitis, or frozen shoulder, is characterized by pain and stiffness due to capsular inflammation and fibrosis. Corticosteroid injections are commonly used but may be contraindicated in some patients. Hyaluronic acid (HA) and ketorolac each have shown benefit, yet evidence on their combined use is limited.

This randomized, double-blind, controlled trial enrolled 56 adults with adhesive capsulitis. Participants were randomized 1:1 to receive either HA plus ketorolac or ketorolac alone as a single intra-articular injection, followed by standardized rehabilitation. Follow-up assessments were conducted at 2, 6, 12, and 24 weeks.

The primary outcome was functional outcome measured by the Thai SPADI. Secondary outcomes included pain (VAS), PROM, analgesic use, and adverse events. Both groups improved significantly in function and pain, without significant between-group differences. However, the HA+ketorolac group showed modest but significant improvements in external rotation and adduction range of motion. Safety outcomes were favorable in both groups, with only one mild adverse event reported.

This study demonstrates that intra-articular HA combined with ketorolac and ketorolac alone are safe and effective alternatives to corticosteroid injection for adhesive capsulitis. The combination may provide additional benefit in range of motion recovery and can be considered in patients for whom corticosteroids are unsuitable.

ELIGIBILITY:
Eligible participants were adults diagnosed with adhesive capsulitis defined by limitation of shoulder motion ≥25 degrees in at least two planes compared to the contralateral side

Inclusion Criteria:

* Adults aged 18-70 years
* Symptom duration of 1-12 months
* Provision of informed consent.

Exclusion Criteria:

* History of trauma or prior surgery to the affected shoulder
* Bilateral adhesive capsulitis
* Uncontrolled diabetes (HbA1C > 7%)
* Abnormal thyroid function
* Prior intra-articular injection in the affected shoulder
* Full-thickness rotator cuff tear on imaging
* History of gastrointestinal bleeding
* Known allergy to hyaluronic acid or NSAIDs
* Systemic conditions affecting joint pain (e.g., SLE, rheumatoid arthritis, osteoarthritis)
* Neurological disorders affecting muscle strength or sensation coagulopathy or bleeding disorders withdrawal or refusal of consent at any time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Shoulder function (Thai SPADI score) | Baseline, 2, 6, 12, and 24 weeks post-injection
  Shoulder Pain and Disability Index (Thai version), patient-reported outcome measure, score range 0-100 (higher score = worse disability)

SECONDARY OUTCOMES:
Pain intensity (VAS score) | Baseline, 2, 6, 12, and 24 weeks post-injection
  Visual Analog Scale for shoulder pain, 0-10 (higher score = worse pain)
Passive range of motion (PROM) | Baseline, 2, 6, 12, and 24 weeks post-injection
  Passive range of motion of the affected shoulder (flexion, extension, abduction, adduction, internal and external rotation) measured with goniometer in degrees
Adverse events | 0-24 weeks post-injection
  Number and type of treatment-related adverse events (mild, moderate, or severe) reported by participants or observed by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Pratantat Charoenchaipong, MD, Principal Investigator — Ramathibodi Hospital; Sorawut Thamyongkit, MD, Study Director — Chakri Naruebodindra Medical Institute
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee SC, Rha DW, Chang WH. Rapid analgesic onset of intra-articular hyaluronic acid with ketorolac in osteoarthritis of the knee. J Back Musculoskelet Rehabil. 2011;24(1):31-8. doi: 10.3233/BMR-2011-0272. PMID 21248398
- [Result] Taheri P, Dehghan F, Mousavi S, Solouki R. Comparison of Subacromial Ketorolac Injection versus Corticosteroid Injection in the Treatment of Shoulder Impingement Syndrome. J Res Pharm Pract. 2017 Oct-Dec;6(4):223-227. doi: 10.4103/jrpp.JRPP_17_57. PMID 29417082
- [Result] Xu J, Qu Y, Li H, Zhu A, Jiang T, Chong Z, Wang B, Shen P, Xie Z. Effect of Intra-articular Ketorolac Versus Corticosteroid Injection for Knee Osteoarthritis: A Retrospective Comparative Study. Orthop J Sports Med. 2020 Apr 10;8(4):2325967120911126. doi: 10.1177/2325967120911126. eCollection 2020 Apr. PMID 32313809
- [Result] Mao B, Peng R, Zhang Z, Zhang K, Li J, Fu W. The Effect of Intra-articular Injection of Hyaluronic Acid in Frozen Shoulder: a Systematic Review and Meta-analysis of Randomized Controlled Trials. J Orthop Surg Res. 2022 Mar 3;17(1):128. doi: 10.1186/s13018-022-03017-4. PMID 35241100
- [Result] Uhm KE, Chang MC. Comparison of Effectiveness of Intraarticular Hyaluronate and Corticosteroid injections in Adhesive Capsulitis: A Systematic Review and Meta-analysis. Pain Physician. 2024 Sep;27(7):387-400. PMID 39353107
- See also: Randomized, double-blind, placebo-controlled trial of 60 patients with adhesive capsulitis. Participants were randomized into four arms (saline, corticosteroid, hyaluronic acid, corticosteroid + hyaluronic acid) — https://pubmed.ncbi.nlm.nih.gov/34766090/